CLINICAL TRIAL: NCT04807894
Title: Prevention of Recurrent Urinary Tract Infection Using Vaginal Testosterone Versus Placebo
Brief Title: Prevention of Recurrent UTI Using Vaginal Testosterone Versus Placebo Placebo
Acronym: PIVoT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Collaborators: American Urological Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 702576
Record Dates: First submitted 2020-10-19; First posted 2021-03-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Urinary Tract Infection; Vaginal Atrophy; Postmenopausal Disorder
Keywords: urinary tract infections,; postmenopausal women; vaginal atrophy,; vaginal flora
MeSH Terms: conditions — Urinary Tract Infections | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaginal Testosterone Cream Arm (Experimental): Women enrolled in this arm will receive vaginal testosterone cream to be applied once each night for two weeks followed by twice-weekly applications for a total duration of nine months.
  Interventions: Drug: Vaginal Cream with Applicator
- Vaginal Placebo Cream Arm (Placebo Comparator): Women enrolled in this arm will receive vaginal placebo cream to be applied once each night for two weeks followed by twice-weekly applications for a total duration of nine months.
  Interventions: Drug: Vaginal Cream with Applicator

INTERVENTIONS:
Drug: Vaginal Cream with Applicator — Vaginal testosterone 300-μg dose will be compounded with 13.5 mg of testosterone propionate in 0.45 mL of polysorbate National Formulary liquid and sufficient emollient cream base to make 45 g total. A calibrated vaginal applicator will be supplied to measure out doses of 1 g each. All study medications will be compounded by a single pharmacy so as to avoid variation in compounding between pharmacies and allow for control of compounding. Randomization will be conducted by the compounding pharmacy to allow for double-blinding of patients and clinicians.
  Other Names: Testosterone Cream

SUMMARY:
Women over the age of 60 years have an estimated 10 to 15 % risk of recurrent urinary tract infections (UTI). This is believed to be due to hormonally induced changes in the vaginal flora associated with menopause. After menopause, there is a chemical changes in the vagina that may predispose to bacterial infections.

The role of vaginal estrogen creams to restore vaginal atrophy and prevent urinary tract infections has been well characterized. Vaginal testosterone (VT) application use in postmenopausal breast cancer patients on aromatase inhibitors have been shown to improve vaginal pH, vaginal atrophy symptom scores, dyspareunia, and vaginal dryness. Although testosterone has been used to improve sexual function in postmenopausal women, the effects of VT on vaginal flora and recurrent UTIs are unknown.

The purpose of this study is to determine whether topically applied vaginal testosterone cream is more effective than placebo in reducing the incidence of urinary tract infections in postmenopausal women with recurrent urinary tract infections and to ascertain the effects of topical estrogen on the vaginal pH and flora.

DETAILED DESCRIPTION:
Background:

Women over the age of 60 years have an estimated 10 to 15 % risk of recurrent urinary tract infections (UTI). This is believed to be due to hormonally induced changes in the vaginal flora associated with menopause. After menopause, there is a chemical changes in the vagina that may predispose to bacterial infections.

The role of vaginal estrogen creams to restore vaginal atrophy and prevent urinary tract infections has been well characterized. Vaginal testosterone (VT) application use in postmenopausal breast cancer patients on aromatase inhibitors have been shown to improve vaginal pH, vaginal atrophy symptom scores, dyspareunia, and vaginal dryness. Although testosterone has been used to improve sexual function in postmenopausal women, the effects of VT on vaginal flora and recurrent UTIs are unknown.

The purpose of this study is to determine whether topically applied vaginal testosterone cream is more effective than placebo in reducing the incidence of urinary tract infections in postmenopausal women with recurrent urinary tract infections and to ascertain the effects of topical estrogen on the vaginal pH and flora.

Methods:

This will be a multi-center randomized, double- blind placebo-controlled study. Participating clinic sites include Maimonides Medical Center and Northwell Health. Subjects will be one hundred postmenopausal women presenting to a gynecology, urogynecology or female urology clinic with a history of three or more microbiologically confirmed symptomatic episodes of urinary tract infection during the either the previous year or two or more within six months.

Patients will randomly assigned to one of two regimens: one group will receive VT cream to be used once each night for two weeks followed by twice-weekly applications for eight months, and the other group will receive a placebo cream to be used in the same manner. Demographic data, vaginal exam including vaginal swab to assess vaginal flora, vaginal pH measurement and vaginal atrophy index measurement will be collected at the initial study visit, again at a study visit at 4.5 months and another at 9 months.

Anticipated Results and Conclusion:

It is anticipated that vaginal testosterone cream will reduce the incidence of urinary tract infections in postmenopausal women when compared to placebo. It is expected that vaginal testosterone will improve vaginal atrophy and flora, thus, decreasing the frequency of urinary tract infections. Future aims of the study will focus on immune-dynamics associated with vaginal testosterone administration.

ELIGIBILITY:
Inclusion Criteria:

* 60-90 yo Female
* Postmenopausal
* Recurrent UTIs (three or more culture confirmed symptomatic episodes of UTI or two or more in the past 6 months).
* English Proficiency
* Unable or unwilling to use topical estrogen.
* Patients with history of or current endometrial or breast cancer and current aromatase inhibitor therapy may also be included in study.
* Patient on oral estrogen therapy may be included.
* Patient with slings, prior vaginal surgery or pessary may be included.

Exclusion Criteria:

* Current UTI/ Dipstick and culture positive (> trace leukocytes or nitrites)
* Antibiotic (vaginal or oral) use in the last 4 weeks
* Current sexually transmitted infection
* Chronic Foley catheter use or chronic ureteral stent placement.
* Vaginal probiotic use in the last 4 weeks
* Patient currently using vaginal estrogen.
* Post-void Residual Volume >150 mL or current diagnosis of urinary retention
* Non-evaluated hematuria (> trace on dipstick, microscopic, gross)
* Unable to complete study tasks or comply with follow up.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is aimed at postmenopausal women with history of recurrent UTIs.
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess whether topical vaginal testosterone cream is more effective than placebo in reducing the incidence of urinary tract infections in postmenopausal women with recurrent urinary tract infections. | 1 month
  Patients will receive months phone calls to assess for symptoms of UTI and urine will be collected in study visits at 1 month to check for presence of UTI.
To assess whether topical vaginal testosterone cream is more effective than placebo in reducing the incidence of urinary tract infections in postmenopausal women with recurrent urinary tract infections. | 4.5 months
  Patients will receive months phone calls to assess for symptoms of UTI and urine will be collected in study visits at 4.5 months to check for presence of UTI.
To assess whether topical vaginal testosterone cream is more effective than placebo in reducing the incidence of urinary tract infections in postmenopausal women with recurrent urinary tract infections. | 9 months
  Patients will receive months phone calls to assess for symptoms of UTI and urine will be collected in study visits at 9 months to check for presence of UTI.
To determine whether topically applied vaginal testosterone cream is more effective than placebo cream in changing vaginal flora and pH in postmenopausal women with recurrent urinary tract infections. | 1 month
  The vaginal pH, vaginal atrophy score, and vaginal swabs for participants will be collected at 1 month to assess whether there is improvement in pH and vaginal atrophy scores as well as normalization of vaginal flora.
To determine whether topically applied vaginal testosterone cream is more effective than placebo cream in changing vaginal flora and pH in postmenopausal women with recurrent urinary tract infections. | 4.5 months
  The vaginal pH, vaginal atrophy score, and vaginal swabs for participants will be collected at 4.5 months to assess whether there is improvement in pH and vaginal atrophy scores as well as normalization of vaginal flora.
To determine whether topically applied vaginal testosterone cream is more effective than placebo cream in changing vaginal flora and pH in postmenopausal women with recurrent urinary tract infections. | 9 months
  The vaginal pH, vaginal atrophy score, and vaginal swabs for participants will be collected at 9 months to assess whether there is improvement in pH and vaginal atrophy scores as well as normalization of vaginal flora.

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No